CLINICAL TRIAL: NCT01852149
Title: Mitralign Percutaneous Annuloplasty First in Man (FIM) Study
Brief Title: Mitralign Percutaneous Annuloplasty First in Man Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitralign, Inc. (Industry)
Collaborators: Medstar Health Research Institute (Other); The Cooper Health System (Other); Cardiovascular Research Center, Brazil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLPR-005
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Functional Mitral Regurgitation
Keywords: Mitral Valve Regurgitation; Coaptation; Mitral Valve Repair; Plication; Leaflet; Annulus; Mitral Annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPAS Implant (Experimental): MPAS Implant
  Interventions: Device: MPAS Implant

INTERVENTIONS:
Device: MPAS Implant — The Mitralign System consists of a set of catheters that enable the physician to position and place sutures and anchors through the posterior (back) annulus of the mitral valve under the guidance of echocardiography and fluoroscopy. Once the anchored sutures are in place, the sutures are pulled together. When the valve leaflets are close together, the sutures are locked with at least one stainless steel lock. The Bident Translation Catheter allows implantation of two pairs of pledgets. Each pair of pledgets plicates the annulus and then the pledgets are locked together from the ventricular side with a lock.
  Other Names: Bident; Plication; Mitral annuloplasty; annulus; Mitral Regurgitation

SUMMARY:
The purpose of this study is to assess the safety and feasibility of the Mitralign Percutaneous Annuloplasty System in humans for the treatment of chronic functional mitral regurgitation. No formal test of hypothesis is proposed for this trial.

DETAILED DESCRIPTION:
The primary objective of this study is to test the ability to safely perform mitral posterior annulus plication with the Mitralign System in eligible patients with chronic functional MR using an endovascular approach. Data obtained from this study, combined with extensive pre-clinical data, will provide important technical and early clinical outcome information that will drive the next phase of clinical investigation and potentially enhance the future design of the Mitralign Percutaneous Annuloplasty System. It is anticipated that the Mitralign System will one day provide physicians with a safe and effective alternative therapy for treating patients who are candidates for mitral valve repair and offer a primary therapy option for patients superior to current treatment modalities.

This is a single-arm, multi-center, prospective study designed to test the safety and feasibility of the MPAS to treat patients with chronic, functional MR by performing plication of the posterior mitral annulus.

Up to a total of 36 patients with chronic functional mitral regurgitation will be enrolled: 1.) Up to 16 patients (12 patients + 1 roll-in patient per site) will be enrolled in Phase I. Up to thirty-four (34) patients will be enrolled in Phase II (MITRALIGN ADVANTAGE). All patients will be followed for 24 months. Up to 5 sites in Europe and South America will participate.

Study procedures include implantation of the MPAS, Trans-Esophogeal Echo, Trans-Thoracic Echo, Blood test, 6-min walk, Quality of Life, Chest X-ray and ECG.

Descriptive Statistics will be conducted for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic functional mitral regurgitation.
* Patient is greater than 18 years old.
* Documented symptoms of CHF - NYHA II-IV.
* Left ventricular ejection fraction between 30 and 60 percent.
* Acceptable candidate for cardiac surgery and/or blood transfusion.
* Patient or legal guardian understands the study requirements and the treatment procedures and provides written Informed Consent before any study- specific tests or procedures are performed.
* Willing to comply with all specified follow-up evaluations.
* Mitral regurgitation grade 2.
* Patient has a mitral plane to apex dimension 5 cm.
* Structurally normal mitral valve.

Exclusion Criteria:

* Patient with significant organic mitral valve pathology such as myxomatous degeneration, mitral valve prolapse or flail leaflets moderate or severe valve calcifications, ruptured papillary muscles or ruptured chordae tendinae.
* Previous mitral valve repair or mitral valve replacement.
* Patient with mitral stenosis.
* Patient with moderate or severe aortic stenosis and or moderate or severe aortic regurgitation.
* Patient with endocarditis.
* MI within 30 days prior to the index procedure.
* Unstable angina.
* Percutaneous Coronary Intervention within 30 days prior to the index procedure.
* CABG within 3 months prior to the index procedure.
* Planned PCI less than 30 days post index procedure.
* Planned CABG within 6 months post index procedure.
* Patient with severe, multivessel coronary artery disease and who cannot tolerate sudden hemodynamic changes or acute hemoglobin drop.
* Cardiogenic Shock characterized by systolic pressure less than 80 mm Hg and or central filling pressure greater than 20 mm Hg, or cardiac index less than 1.8 liters per minute per m2 or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure greater than 80 mm Hg and a cardiac index greater than 1.8 liters per minute per m2.
* Patient with peripheral vascular disease or tortuousity that would prevent percutaneous access with a 14 Fr introducer sheath or intervention with the Mitralign system.
* Cerebrovascular Accident within the past 6 months.
* Acute or chronic renal dysfunction creatinine greater than 2.0mg per dl or 177µmolper dl
* Anemia Hb greater than 10 g per dl.
* Thrombocytopenia platelet count less than 100,000 per mm3) or thrombocytosis platelet greater than 750,000 per mm3).
* Bleeding disorders or hypercoaguable state.
* Active peptic ulcer or active gastrointestinal bleeding.
* Contraindication to therapy with antiplatelet or anticoagulant drugs.
* Contraindications to or patient's refusal of blood transfusions.
* Known allergy to stainless steel or platinum iridium or polyester.
* Any prior true anaphylactic reaction to contrast agents defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure.
* Pregnancy or female of childbearing potential with a positive pregnancy test within 24 hours before the index procedure or undergoing any angiography or x-ray, or lactating.
* Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
* Life expectancy of less than 24 months due to other medical condition.
* Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.
* Patient with impaired judgment.
* Patient having to undergo emergency treatment.
* Thrombus in left ventricle or left atrium.
* Echocardiographic evidence of congenital, pericardial or infiltrative heart disease.
* Suboptimal echocardiographic (TTE) windows, leading to incomplete quantification of FMR or anatomic assessment.
* Significant subvalvular trabecularization, muscle bridges and pockets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint will assess acute safety defined as the incidence of Device-related NACE (net adverse clinical events which includes Device Related Mortality, MI, Cardiac Tamponade and stroke) at 30 days | 30 Days post implant
  The primary study endpoint will assess acute safety using a composite clinical endpoint of device-related net adverse cardiac events (NACE) at 30 days. The components of NACE are defined as the occurrence of device related mortality, myocardial infarction, cardiac tamponade, cardiac surgery or stroke in per protocol population

SECONDARY OUTCOMES:
Echocardiographic measures | 6 Months
  Measurement of Ventricular diameter and Mitral Regurgitant Grade

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Principal Investigator — Universitats Klinikum Bonn; Kimberlie O'Connell, MBA, Study Director — Mitralign, Inc.
Locations (5):
- Instituto Dante Passanese de Cardiologia, São Paulo, Brazil
- Germany (3):
  - Universitats Klinikum Bonn, Bonn
  - Elisabeth-Krankenhaus Essen, Essen
  - Asklepios Klinik St Georg, Hamburg
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Nickenig G, Schueler R, Dager A, Martinez Clark P, Abizaid A, Siminiak T, Buszman P, Demkow M, Ebner A, Asch FM, Hammerstingl C. Treatment of Chronic Functional Mitral Valve Regurgitation With a Percutaneous Annuloplasty System. J Am Coll Cardiol. 2016 Jun 28;67(25):2927-36. doi: 10.1016/j.jacc.2016.03.591. PMID 27339489
- See also: Sponsor website — http://www.mitralign.com